## NASAL SWAB COLLECTION CONSENT FORM

As-salamua-likum, sir. My name is \${enumname}. I am working for Innovations for Poverty Action (IPA) - a non-profit organization. In collaboration with Bangladesh Government's Access to Information (A2i), Yale University and Stanford University, we are conducting research to understand how to reduce infectious disease in your community.

We would like to swab the nose of the person in your household who spends the most time outside the house to determine if they are infected with coronavirus. Measuring the number of people getting infected will help us understand if the policies in the study are being able to control the spread of COVID-19. We will come back 3 more times over the next 1-2 months. To compensate you for your time, we're providing 40 taka. Unfortunately, we won't be able to provide the results of the test for 6-12 months because we have so many samples to process.

Which adult household member leaves the bari most often to go to public places, such as the mosque, markets, tea stalls, restaurants, or political or religious events?

Response: Record hh member's name

b. Don't want to be bothered

Is \_\_[name of person who spends the most time out of the house]\_\_\_\_ here?

If the person is NOT present and has consented, say the following:

Do you think \_\_\_ [name of person who spends the most time out of the house]\_\_\_\_ would be willing to swab his/her nose?

If yes, record "other person reported likely to consent"

- Thank you for your time. What time will \_\_\_ [name of person who spends the most time out of the house]\_\_\_\_ be home later today?

- What time will \_\_\_ [name of person who spends the most time out of the house]\_\_\_\_ be home tomorrow so we can ask for his/her consent?

If no, record "other person reported not likely to consent"

- Why do you think \_\_\_ [name of person who spends the most time out of the house]\_\_\_\_ would not want to swab his/her nose?

A. Don't want to swab the nose

You can swab your nose on your own. You

simple insert the swab into the tip of your

It's a very simple procedure. You don't have

hostile and turn it 4 times.

| | to put the swab very far into your nose or into your throat. |
|---|---|
| c. It will hurt | It is very simple and will not hurt. You can do it by yourself or a trained professional can help you. |
| d. Time-consuming | It will take just 1 minute to swab your nose. |
| e. Don't want to know | Your participation will help us learn how the spread of infectious diseases can be reduced and that learning might help the government and NGOs to fight the current and the future pandemics to improve your community's health and wellbeing. We won't be able to tell you your results because the lab has many samples to process and it will take 6-12 months to process al of the samples |

 Do you still think that \_\_\_\_[name of person who spends the most time out of the house]\_\_\_\_ would not want to swab his/her nose?

If the person is present and has indicated they would consent, say the following:

We will determine whether you have been exposed to coronavirus by swabbing your nose. We will test the swab for coronavirus. We may also ask you a few questions about your health and vaccination status and ask you or your family members 5-10 minutes of questions about who you interacted with yesterday. Your answers will be anonymously combined with the answers of other people in your community and people from many other communities. We will use the responses to inform organizations such as the government, BRAC, and healthcare providers how to best protect you and your community.

There is minimal physical risk to you from swabbing your nose. You may feel temporary discomfort, and there is a very small chance that your nose may bleed.

This is a research study so we do not provide healthcare. However, your participation will help us learn how the spread of infectious diseases can be reduced and that learning might help the government and NGOs to fight the current and the future pandemics.

The results from your test will strictly remain confidential and protected and will only be used for research purposes. They will never be shared with your neighbors or the community or with anyone outside of the research teams from IPA and Yale. We will

only analyze the test results at the community level and will not provide you or anyone else with your individual test results.

Participation is voluntary and you can withdraw your participation anytime or refuse to participate. Refusal to participate will not result in any penalty or loss of existing benefits.

Your information or biospecimens collected as part of the research will not be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you or your legally authorized representative.

Do you have any questions about the test we would like to conduct?

If you have a question later, or if you have concerns or complaints about this interview, please contact Asraul Houqe Khan (Eitu), Sr. Data Management Coordinator, Innovations for Poverty Action (IPA) Bangladesh. Phone: (+880)1716 590539. You can also share your concerns or complaints with the Bangladesh Medical Research Council by contacting info@bmrcbd.org.

Are you willing to swab your nose or have someone help you swab your nose?